CLINICAL TRIAL: NCT00006124
Title: Phase IIb/III Chemoprevention Trial of Celecoxib to Prevent Recurrence of Superficial Bladder Cancer
Brief Title: Celecoxib in Treating Patients With Bladder Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2009-00869; ID99-368; N01CN85186 (Other Grant/Funding Number: US NIH Grant/Contract Award Number)
Record Dates: First submitted 2000-08-03; First posted 2003-01-27 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (celecoxib) (Experimental): Patients receive oral celecoxib twice daily.
  Interventions: Drug: celecoxib
- Arm II (placebo) (Placebo Comparator): Patients receive oral placebo twice daily.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: celecoxib — Given orally
  Other Names: Celebrex; SC-58635
  Arms: Arm I (celecoxib)
Drug: placebo — Given orally
  Other Names: PLCB
  Arms: Arm II (placebo)

SUMMARY:
This randomized phase IIb/III trial is studying celecoxib to see how well it works in preventing disease recurrence in patients who have bladder cancer. Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of celecoxib may be an effective way to prevent the recurrence of bladder cancer

DETAILED DESCRIPTION:
OBJECTIVES:

I. Compare the time to recurrence after treatment with celecoxib vs placebo in patients with superficial transitional cell carcinoma of the bladder at high risk for recurrence.

II. Correlate the modulation of one or more biomarkers with recurrence of bladder cancer and confirm the value of the marker(s) as a surrogate endpoint biomarker for bladder cancer and celecoxib.

III. Determine the toxicity of celecoxib in these patients. IV. Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to center and presence of Tis disease (yes vs no). Patients are randomized to one of two arms.

Arm I: Patients receive oral celecoxib twice daily.

Arm II: Patients receive oral placebo twice daily.

Treatment continues in both arms for 1-2 years in the absence of unacceptable toxicity, development of recurrent or invasive bladder carcinoma, or development of a second malignancy requiring radiotherapy or systemic therapy.

Quality of life is assessed at baseline and at week 54.

Patients are followed at 6 weeks and then every 12 weeks until the last randomized patient has been on the study for 1 year or until disease recurrence.

ELIGIBILITY:
Criteria:

* No concurrent radiotherapy
* No prior angioplasty
* No concurrent chemotherapy
* No concurrent oral or IV corticosteroids for more than 2 consecutive weeks or orally inhaled corticosteroids for more than 4 consecutive weeks during any 6 month period of the study
* Chronic nasally inhaled steroids allowed provided patient agrees to use mometasone or, in countries where mometasone is not available, fluticasone
* No prior coronary bypass surgery
* At least 30 days since prior investigational medication
* No other prior malignancy within the past 5 years except:
* No prior pelvic radiotherapy
* Histologically proven superficial transitional cell carcinoma of the bladder at high risk for recurrence, meeting 1 of the following staging criteria:
* Stage Ta (grade 3 OR multifocal OR at least 2 occurrences, including current tumor, within the past 12 months)
* Stage T1 (any grade)
* Stage Tis
* Patients with Ta or T1 lesions must have undergone complete transurethral resection of bladder tumor within the past 9 months
* No carcinoma involving the prostatic urethra or upper urinary tract
* Must have received the following prior to randomization:
* Induction course of BCG comprising 6 weekly intravesical doses (at least 4 doses if BCG intolerant)
* Additional induction courses of BCG allowed
* Maintenance course of BCG comprising 3 weekly doses (at least 1 dose if BCG intolerant)
* No evidence of disease by cystoscopy (with or without biopsy) and bladder cytology prior to initiation of maintenance BCG
* Concurrent interferon allowed
* Zubrod 0-2 or ECOG 0-2
* WBC at least 3,000/mm^3
* Hemoglobin at least lower limit of normal
* Platelet count at least 125,000/Mm^3
* No significant bleeding disorder
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT and SGPT no greater than 1.5 times ULN
* No chronic or acute hepatic disorder
* Creatinine no greater than 1.5 times ULN
* No chronic or acute renal disorder
* Normal kidneys and ureters on imaging study within the past 9 months
* No active inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis)
* No active pancreatitis
* No esophageal, gastric, pyloric channel, or duodenal ulceration that was diagnosed or treated within the past 30 days
* No history of cardiovascular disease, including any of the following conditions:
* Stroke
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other medical or psychological condition that would preclude study participation
* No hypersensitivity or adverse reactions to sulfonamides, cyclooxygenase (COX)-2 inhibitors, salicylates, or other NSAIDs
* Nonmelanomatous skin cancer cured by excision
* Carcinoma in situ of the cervix
* Stage 0 chronic lymphocytic leukemia
* Other malignancy for which patient has no current evidence of disease, has received no therapy within the past 6 months, has no concurrent or planned therapy, and has an expected disease-free survival of at least 5 years
* No concurrent immunotherapy
* At least 2 weeks since prior aspirin or nonsteroidal anti-inflammatory drugs (NSAIDs) except cardioprotective dose (no greater than 100 mg/day) of aspirin
* No concurrent chronic NSAIDs except oral cardioprotective dose (no greater than 100 mg/day) of aspirin
* Concurrent chronic use is defined as a frequency of at least 3 times per week for more than 2 consecutive weeks per year
* No other concurrent investigational drug
* No other concurrent systemic therapy
* No concurrent lithium or fluconazole
* No other concurrent hormonal therapy except hormone replacement (i.e., estrogen or thyroid hormone replacement)
* Myocardial infarction
* Angina
* Congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2000-06; Primary Completion 2006-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Time to recurrence | 3 years

SECONDARY OUTCOMES:
Modulation of biomarkers | 3 years
Correlation of biomarkers with tumor recurrence | 3 years
Adverse events as measured by NCI CTC v2.0 | 3 years
Quality of life as measured by EORTC QLQ-C30 v3.0 | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Anita Sabichi, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States